CLINICAL TRIAL: NCT00004471
Title: Phase I Pilot Study of Gene Therapy for Cystic Fibrosis Using Cationic Liposome Mediated Gene Transfer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Purpose: Treatment
Other Study IDs: 199/13941; UAB-6097; UAB-F930923001
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Cystic Fibrosis
Keywords: cardiovascular and respiratory diseases; cystic fibrosis; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — Cystic Fibrosis; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases

INTERVENTIONS:
Genetic: pGT-1 gene lipid complex

SUMMARY:
OBJECTIVES:

Determine whether copies of the cystic fibrosis gene (pGT-1) can be delivered to the cells lining the nose of cystic fibrosis patients using cationic liposome (DMRIE/DOPE) mediated gene transfer.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Under direct visualization, patients receive lipid/DNA formulation (pGT-1 lipid complex) by syringe instillation over 30 minutes to the right inferior nasal turbinate.

Patients are followed daily for 7 days, twice a week for 3 weeks, every 2-3 weeks for 10 weeks, then every 3 months thereafter.

ELIGIBILITY:
* Cystic fibrosis patients
* Not pregnant Fertile patients must use effective contraception

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9
Dates: Start 1995-08; Primary Completion 2001-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Sorscher, Study Chair — University of Alabama at Birmingham